CLINICAL TRIAL: NCT03717194
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group, to Evaluate the Effect of Ertugliflozin on Cardiac Function in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control and Stage B Heart Failure
Brief Title: Effect of Ertugliflozin on Cardiac Function in Diabetes
Acronym: ERTU-GLS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Soo Lim (Other)
Collaborators: MSD Korea Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Organization: Seoul National University Bundang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-2018-498-002
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Type2 Diabetes; Heart Failure
Keywords: type 2 diabetes; heart failure; ertugliflozin; Global longitudinal strain (GLS)
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2 | interventions — ertugliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ertugliflozin (Experimental): Ertugliflozin 5 mg in addition to their preexisting metformin and/or DPP4 inhibitor
  Interventions: Drug: Ertugliflozin
- Control group (Placebo Comparator): Placebo in addition to their preexisting metformin and/or DPP4 inhibitor
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ertugliflozin — Ertugliflozin as add-on to Metformin and/or DPP4 inhibitors in patients with inadequately controlled type 2 diabetes
  Other Names: Steglatro
  Arms: Ertugliflozin
Drug: Placebo — Placebo as add-on to Metformin and/or DPP4 inhibitors in patients with inadequately controlled type 2 diabetes
  Arms: Control group

SUMMARY:
The aim of this study is to investigate the beneficial role of ertugliflozin, a new SGLT2 inhibitor, in cardiac function via measuring GLS as well as other hemodynamic factors using echocardiogram in patients with T2D and HF, who are not controlled with oral antidiabetic medications including DPP4 inhibitors.

DETAILED DESCRIPTION:
This study is a phase 3, randomized, double-blind, active-competitor, parallel-group study that is anticipated to enroll 120 patients. Patients taking metformin and/or DPP4 inhibitors as per local label for ≥12 weeks without a dose adjustment before enrollment will be eligible for screening. All patients will have a screening period comprised of an up to 2-week screening phase prior to randomization. In order to qualify for randomization, patients must demonstrate compliance based upon pill count (80%) and discretion of the investigators during the Run-in phase.

Glycated hemoglobin (HbA1c) and fasting plasma glucose (FPG) will be masked to patients after randomization. To prevent partial unblinding, urinary glucose excretion (UGE) results will be masked to patients. Urine glucose, albumin, calcium, and creatinine will be measured separately on-site visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2D taking oral antidiabetic medications (metformin and/or DPP4 inhibitors) except SGLT2 inhibitors for at least 12 weeks without a dose adjustment before enrollment.
* eGFR ≥ 45 mL/min/1.73 m2.
* Stage B HF identified on the basis of either structural or functional markers.

Exclusion Criteria:

* Type 1 diabetes mellitus
* At the time of screening age <20 years
* HbA1c <7% or HbA1c >9.5% at Screening
* FPG >15 mmol/L (270 mg/dL) measured by the laboratory at Screening (Visit 1), and confirmed (>15 mmol/L [>270 mg/dL]) by a repeat test before randomization
* Treated with insulin and/or GLP-1R agonist within 12 weeks preceding the Screening Visit.
* Women of childbearing potential with no effective contraceptive method
* History of gastric surgery including history of gastric banding within 3 years before the Screening Visit
* History of diabetic ketoacidosis or nonketotic hyperosmolar coma prior to the Screening Visit
* Mean blood pressure after 3 separate measurements >180 mmHg in systolic blood pressure (SBP) or >95 mmHg in diastolic blood pressure (DBP)
* Patients with current or prior symptoms of HF.
* Patients with severe anemia, severe respiratory, hepatic, neurological, psychiatric disorders or active malignant tumor or other major systemic disease or patients with short life expectancy making implementation of the protocol or interpretation of the study results difficult
* Aspartate aminotransferase and/or alanine aminotransferase: >3 times the upper limit of the normal laboratory range (ULN)
* Total bilirubin: >1.5 times ULN (except in case of Gilbert's syndrome)
* Use of systemic glucocorticoids (excluding topical or ophthalmic, application or inhaled forms) for more than 10 consecutive days within 90 days prior to the Screening Visit
* Patient who has taken other investigational drugs or prohibited therapy for this study within 3 months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospita;, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Background] Neal B, Perkovic V, Matthews DR. Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes. N Engl J Med. 2017 Nov 23;377(21):2099. doi: 10.1056/NEJMc1712572. No abstract available. PMID 29166232
- [Background] Krishnasamy R, Isbel NM, Hawley CM, Pascoe EM, Burrage M, Leano R, Haluska BA, Marwick TH, Stanton T. Left Ventricular Global Longitudinal Strain (GLS) Is a Superior Predictor of All-Cause and Cardiovascular Mortality When Compared to Ejection Fraction in Advanced Chronic Kidney Disease. PLoS One. 2015 May 15;10(5):e0127044. doi: 10.1371/journal.pone.0127044. eCollection 2015. PMID 25978372
- [Background] Hunt SA, Baker DW, Chin MH, Cinquegrani MP, Feldman AM, Francis GS, Ganiats TG, Goldstein S, Gregoratos G, Jessup ML, Noble RJ, Packer M, Silver MA, Stevenson LW, Gibbons RJ, Antman EM, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Jacobs AK, Hiratzka LF, Russell RO, Smith SC; American College of Cardiology; American Heart Association. ACC/AHA guidelines for the evaluation and management of chronic heart failure in the adult: executive summary. J Heart Lung Transplant. 2002 Feb;21(2):189-203. doi: 10.1016/s1053-2498(01)00776-8. No abstract available. PMID 11834347
- [Background] Kosmala W, Jellis CL, Marwick TH. Exercise limitation associated with asymptomatic left ventricular impairment: analogy with stage B heart failure. J Am Coll Cardiol. 2015 Jan 27;65(3):257-66. doi: 10.1016/j.jacc.2014.10.044. Epub 2014 Dec 19. PMID 25533754
- [Background] Kramer DG, Trikalinos TA, Kent DM, Antonopoulos GV, Konstam MA, Udelson JE. Quantitative evaluation of drug or device effects on ventricular remodeling as predictors of therapeutic effects on mortality in patients with heart failure and reduced ejection fraction: a meta-analytic approach. J Am Coll Cardiol. 2010 Jul 27;56(5):392-406. doi: 10.1016/j.jacc.2010.05.011. PMID 20650361
- [Background] Devereux RB, Alonso DR, Lutas EM, Gottlieb GJ, Campo E, Sachs I, Reichek N. Echocardiographic assessment of left ventricular hypertrophy: comparison to necropsy findings. Am J Cardiol. 1986 Feb 15;57(6):450-8. doi: 10.1016/0002-9149(86)90771-x. PMID 2936235
- [Background] Lang RM, Bierig M, Devereux RB, Flachskampf FA, Foster E, Pellikka PA, Picard MH, Roman MJ, Seward J, Shanewise JS, Solomon SD, Spencer KT, Sutton MS, Stewart WJ; Chamber Quantification Writing Group; American Society of Echocardiography's Guidelines and Standards Committee; European Association of Echocardiography. Recommendations for chamber quantification: a report from the American Society of Echocardiography's Guidelines and Standards Committee and the Chamber Quantification Writing Group, developed in conjunction with the European Association of Echocardiography, a branch of the European Society of Cardiology. J Am Soc Echocardiogr. 2005 Dec;18(12):1440-63. doi: 10.1016/j.echo.2005.10.005. No abstract available. PMID 16376782
- [Background] Nagueh SF, Appleton CP, Gillebert TC, Marino PN, Oh JK, Smiseth OA, Waggoner AD, Flachskampf FA, Pellikka PA, Evangelista A. Recommendations for the evaluation of left ventricular diastolic function by echocardiography. J Am Soc Echocardiogr. 2009 Feb;22(2):107-33. doi: 10.1016/j.echo.2008.11.023. No abstract available. PMID 19187853
- [Background] Reisner SA, Lysyansky P, Agmon Y, Mutlak D, Lessick J, Friedman Z. Global longitudinal strain: a novel index of left ventricular systolic function. J Am Soc Echocardiogr. 2004 Jun;17(6):630-3. doi: 10.1016/j.echo.2004.02.011. PMID 15163933
- [Background] Lima MSM, Villarraga HR, Abduch MCD, Lima MF, Cruz CBBV, Sbano JCN, Voos MC, Mathias W Junior, Tsutsui JM. Global Longitudinal Strain or Left Ventricular Twist and Torsion? Which Correlates Best with Ejection Fraction? Arq Bras Cardiol. 2017 Jul;109(1):23-29. doi: 10.5935/abc.20170085. Epub 2017 Jun 29. PMID 28678927
- [Background] Medvedofsky D, Kebed K, Laffin L, Stone J, Addetia K, Lang RM, Mor-Avi V. Reproducibility and experience dependence of echocardiographic indices of left ventricular function: Side-by-side comparison of global longitudinal strain and ejection fraction. Echocardiography. 2017 Mar;34(3):365-370. doi: 10.1111/echo.13446. Epub 2017 Feb 9. PMID 28185312
- [Derived] Lim S, Bae JH, Oh H, Hwang IC, Yoon YE, Cho GY. Effect of ertugliflozin on left ventricular function in type 2 diabetes and pre-heart failure: the Ertu-GLS randomized clinical trial. Cardiovasc Diabetol. 2024 Oct 22;23(1):373. doi: 10.1186/s12933-024-02463-0. PMID 39438942

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Ertugliflozin 5 mg once daily
- Control Group: Placebo once daily
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 51 | 51
Completed | 48 | 46
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.9) | 65.3 (8.4) | 63.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 39
  Male | 34 | 29 | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 26.3 (2.9) | 26.4 (3.6) | 26.4 (2.9)
Glycated hemoglobin [Mean (Standard Deviation); unit: %] | 8.3 (1.0) | 8.4 (1.1) | 8.4 (1.1)
Estimated glomerular filtration rate [Mean (Standard Deviation); unit: mL/min/1.73 m2] | 90.1 (17.6) | 86.9 (16.8) | 88.5 (17.3)
Hypertension [Number; unit: participants] | 35 | 35 | 70
Dyslipidemia [Number; unit: participants] | 48 | 41 | 89

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Global Longitudinal Strain (LVGLS)
Description: Change in LVGLS after 24 weeks of treatment
Time Frame: Baseline, Week 24
Measure: Mean (Standard Deviation); unit: % of LVGLS
Groups:
- Ertugliflozin Group: Ertugliflozin 5 mg in addition to their preexisting oral antidiabetic medications, except for other SGLT2 inhibitors, or insulin
- Control Group: Placebo in addition to their preexisting oral antidiabetic medications, except for other SGLT2 inhibitors, or insulin
Arm/Group | Ertugliflozin Group | Control Group
Number analyzed (Participants) | 51 | 51
% of LVGLS | 16.6 (2.8) | 16.4 (2.6)

2. Secondary Outcome: Left Ventricular Mass Index (LVMI)
Description: Change in LVMI after 24 weeks of treatment
Time Frame: Baseline, Week 24
Measure: Mean (Standard Deviation); unit: g/m2
Arm/Group | Ertugliflozin Group | Control Group
Number analyzed (Participants) | 51 | 51
g/m2 | 92.6 (22.7) | 99.1 (22.5)

3. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Change in LVEF after 24 weeks of treatment
Time Frame: Baseline, Week 24
Measure: Mean (Standard Deviation); unit: % of LVEF
Arm/Group | Ertugliflozin Group | Control Group
Number analyzed (Participants) | 51 | 51
% of LVEF | 61.3 (7.0) | 61.5 (5.9)

4. Secondary Outcome: E/e' Ratio
Description: Change in E/e' ratio after 24 weeks of treatment
Time Frame: Baseline, Week 24
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Ertugliflozin Group | Control Group
Number analyzed (Participants) | 51 | 51
ratio | 10.6 (3.1) | 10.4 (2.9)

5. Secondary Outcome: Left Atrium Ventricular Index (LAVI)
Description: Change in LVVI after 24 weeks of treatment
Time Frame: Baseline, Week 24
Measure: Mean (Standard Deviation); unit: mL/m2
Arm/Group | Ertugliflozin Group | Control Group
Number analyzed (Participants) | 51 | 51
mL/m2 | 35.5 (11.3) | 35.3 (11.1)

6. Secondary Outcome: Left Ventricular End-diastolic Volume (LVEDV)
Description: Change in LVEDV after 24 weeks of treatment
Time Frame: Baseline, Week 24
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ertugliflozin Group | Control Group
Number analyzed (Participants) | 51 | 51
mL | 82.2 (24.7) | 75.0 (17.8)

7. Other Pre Specified Outcome: N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP)
Time Frame: Baseline, Week 24
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Troponin-T
Time Frame: Baseline, Week 24
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Angiotensin-converting Enzyme 2 (ACE2)
Time Frame: Baseline, Week 24
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Angiotensin (1-7)
Time Frame: Baseline, Week 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Over a 24-week period
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 6/51 | 5/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (N=51) | Control Group (N=51)
Hypoglycemia (Endocrine disorders) | 3 | 1
Genital infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 3
Dehydration (Endocrine disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT03717194/Prot_SAP_000.pdf